CLINICAL TRIAL: NCT00299039
Title: A Randomized Controlled Trial Comparing Combination Therapy of Acetaminophen Plus Ibuprofen Versus Tylenol #3® for the Treatment of Pain After Breast Surgery.
Brief Title: T3AI-Pain After Breast Surgery
Acronym: T3AI
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Nova Scotia Health Authority (Other)
Responsible Party: Dr. Alex Mitchell, Dalhousie University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CDHA008
Record Dates: First submitted 2006-03-02; First posted 2006-03-06 (Estimated); Last update posted 2009-02-02 (Estimated); Status verified 2008-09

CONDITIONS: Pain; Breast Diseases
Keywords: Randomized controlled trial; Clinical trial; Breast tumor surgery; Outpatient surgery; Analgesia; Outpatient analgesia; Post surgical analgesia; ≥ 18 and ≤ 70 years of age; Elective outpatient breast surgery for:; lumpectomy/quadrantectomy +/- Sentinel Lymph Node Biopsy; lumpectomy/quadrantectomy with Axillary Node Dissection; simple mastectomy +/- Sentinel Lymph Node Biopsy; Modified Radical mastectomy
MeSH Terms: conditions — Pain; Breast Diseases; Agnosia | interventions — Acetaminophen; Codeine; Ibuprofen

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- 1 (Active Comparator)
  Interventions: Drug: acetaminophen plus codeine
- 2 (Active Comparator)
  Interventions: Drug: acetaminophen plus ibuprofen

INTERVENTIONS:
Drug: acetaminophen plus codeine — capsules four times daily until pain free or for a maximum of seven days
  Arms: 1
Drug: acetaminophen plus ibuprofen — capsules four times daily until pain free or for a maximum of seven days
  Arms: 2

SUMMARY:
Current standard of care for post-operative analgesia after breast surgery in CDHA is Tylenol #3® (300 mg acetaminophen, 30 mg codeine, 15 mg caffeine per tablet). We are proposing to test the analgesic efficacy of acetaminophen plus ibuprofen against Tylenol #3® in patients undergoing outpatient breast surgery.

DETAILED DESCRIPTION:
Block randomization will be used to randomize patients to one of two combinations. Group A will receive capsules containing 650 mg Acetaminophen plus 400 mg Ibuprofen. Group B will receive capsules containing 600 mg Acetaminophen, 15 mg caffeine and 60 mg codeine. Capsules are placed in identical dossettes containing a seven day supply. Patients are instructed to start taking their medications post-op and continue until they are pain free. All participants are given a series of blank Visual Analogue scales and Likert scales and instructed to record their level of pain intensity and pain relief four times per day for the entire week. Peri-operative pain management will be standardized. Patients will not receive pre-operative analgesics. Intra-operative analgesia will be intravenous opioids as selected by anaesthesiology. No local/regional anaesthesia will be used. Intravenous ketorolac will not be allowed for trial participants. All patients will receive intravenous opioid and anti-emetic if required in PACU. Any patients with peri-operative complications or other problems requiring admission or alternative analgesics will be excluded.

ELIGIBILITY:
Inclusion Criteria:

* ages 18 to 70 inclusive
* outpatient breast surgery: lumpectomy; mastectomy, simple or modified; with or without sentinel lymph node biopsy, axillary node dissection.

Exclusion Criteria:

* allergies to acetaminophen, NSAIDs, ASA or codeine.
* asthma.
* recent reported history of upper GI bleeding.
* daily analgesic use (OTC or opioid) pre-operatively.
* any opioid use in the week prior to surgery.
* reported history of PUD if not on PPI regularly.
* anticoagulant use (low dose ASA excepted).
* renal disease or impairment.
* reported history of liver disease.
* pregnancy.
* major operative complications.
* patients requiring admission.
* communication barrier.
* cognitive or memory impairment.
* reported history of drug and/or alcohol abuse.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2006-05; Primary Completion 2008-06 (Actual); Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
VAS Scores. | mean and daily
maximum VAS scores. | daily
Likert scores. | mean daily and final
Patient satisfaction with analgesic regimen. | day 7
Treatment failures-inadequate pain relief or inability to tolerate side effects. | daily
Time to stopping medication. | day 7

SECONDARY OUTCOMES:
Total Pain relief (TOTPAR). | daily
Sum of pain intensity differences (SPID). | day7
Amount of medication used. | day 7
Incidence of side effects. | day 7
Compliance with regimen. | day 7

CONTACTS AND LOCATIONS:
Overall Officials: Alex D Mitchell, MD, Principal Investigator — CDHA, Dalhousie University
Locations (1):
- QEII Health Sciences Centre, Halifax, Nova Scotia, Canada